CLINICAL TRIAL: NCT01955187
Title: European Multicenter and Open-Label Controlled Randomized Trial to Evaluate the Efficacy of Sequential Treatment With Tacrolimus-Rituximab Versus Steroids Plus Cyclophosphamide in Patients With Primary Membranous Nephropathy (The STARMEN Study)
Brief Title: Sequential Therapy With Tacrolimus and Rituximab in Primary Membranous Nephropathy
Acronym: STARMEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Hospital Universitario Fundación Alcorcón (Other); Fundación para la Investigación Biomédica Hospital Universitario 12 de Octubre (Unknown); Biobanco REDinREN (Unknown); ERA-EDTA (Unknown); REDinREN (Unknown); Spanish Society of Nephrology (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); University Hospital, Aachen (Other)
Responsible Party: Principal Investigator, Manel Praga, MD, MD, PhD, Hospital Universitario 12 de Octubre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STARMEN 01-2013; 2013-000226-55 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2013-10-07 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: MEMBRANOUS NEPHROPATHY
Keywords: SEQUENTIAL THERAPY; PRIMARY MEMBRANOUS NEPHROPATHY; TACROLIMUS; RITUXIMAB
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Tacrolimus; Rituximab; Methylprednisolone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential therapy: Tacrolimus-Rituximab (Experimental): Tacrolimus: Initial dose of 0.05 mg/Kg/day PO, adjusted to blood levels (5- 7 ng/ml) for six months. Starting at the end of month 6, tacrolimus will be reduced by 25% per month, resulting in a complete withdrawal at the end of month 9.
  Interventions: Drug: TACROLIMUS; Drug: RITUXIMAB
- Cyclical therapy: Corticosteroids and Cyclophosphamide (Active Comparator): Month 1, 3 and 5: 1g IV methylprednisolone daily for three doses, oral methylprednisolone (0.5mg/kg/day) Month 2, 4 and 6: Oral Cyclophosphamide (2.0 mg/kg/day)
  Interventions: Drug: METHYLPREDNISOLONE; Drug: CYCLOPHOSPHAMIDE

INTERVENTIONS:
Drug: TACROLIMUS — Initial dose: 0.05 mg/Kg/day, adjusted to achieve blood trough levels of 5-7 ng/ml) for six months. Starting at the end of month 6, tacrolimus dosage will be reduced by 25% per month, resulting in a complete withdrawal at the end of month 9.
  Other Names: TACROLIMUS, ADVAGRAF
  Arms: Sequential therapy: Tacrolimus-Rituximab
Drug: RITUXIMAB — A dose 1 g IV will be given during month 6 (at day 180), before the onset of tacrolimus dose reduction
  Other Names: RITUXIMAB, MABTHERA
  Arms: Sequential therapy: Tacrolimus-Rituximab
Drug: METHYLPREDNISOLONE — Month 1: 1g IV methylprednisolone daily for three doses (days 1, 2, and 3), Oral methylprednisolone (0.5mg/kg/day) for 27 days (days 4 to 30). Months 3, and 5: Repeat Month 1.
  Other Names: METHYLPREDNISOLONE, URBASON, SOLUMODERIN
  Arms: Cyclical therapy: Corticosteroids and Cyclophosphamide
Drug: CYCLOPHOSPHAMIDE — Month 2: Oral Cyclophosphamide (2.0 mg/kg/day) for 30 days. Months 4, and 6: Repeat month 2.
  Other Names: CYCLOPHOSPHAMIDE, GENOXAL
  Arms: Cyclical therapy: Corticosteroids and Cyclophosphamide

SUMMARY:
In this study, investigators will evaluated the long-term efficacy and safety (two years) of Tacrolimus-Rituximab (RTX) therapy compared to Methylprednisolone-Cyclophosphamide (CYC) therapy in patients with primary Membranous Nephropathy (MN).

PRINCIPAL OBJECTIVE To evaluate whether sequential therapy with tacrolimus leads to a greater increase in the proportion of primary MN patients with Complete or Partial Remission when compared with patients receiving standard treatment. It will be assessed 24 months after the beginning of treatment.

Phase of the trial: and design: Phase III study, open label, randomized, and active controlled trial.

This study will have 3 stages: screening and recruitment of patients for 18 months, treatment period for six months in corticosteroids plus CYC group and 9 months in Tacrolimus-RTX group, and finally post-treatment follow-up period until to complete 24 months of follow-up since initial treatment.

This study will compare the standard therapy for primary MN patients with nephrotic range proteinuria (active control of steroids plus CYC) with a novel sequential therapy of tacrolimus and RTX, an approach of potential high efficacy, low toxicity and more acceptable safety profile.

DETAILED DESCRIPTION:
PRIMARY AND SECONDARY ENDPOINTS/OUTCOME MEASURES

Primary end-point:

The proportion of patients reaching CR defined as a reduction of proteinuria since baseline level to a value equal or lower than 0.5 g/24 h proteinuria plus stable renal function (eGFR ≥ 45 ml/min/1.73m2) or PR defined as a reduction of proteinuria since baseline level to a value less than 3.5 g/24 h and 50% lower than baseline proteinuria plus stable renal function (eGFR ≥ 45ml/min/1.73m2) at 24 months of study treatment.

Secondary end-points

* The proportion of patients with Limited response (LR) defined as a reduction of proteinuria since baseline level > 50% but to a value > 3.5g/24 h. at 12, 18 and 24 months of study treatment..
* The number of patients with an increase ≥ 50% of serum creatinine (SCr) from baseline at 12, 18 and 24 months (end of the follow-up).
* The time of renal survival (status free of increase ≥ 50% of baseline SCr) in both arms overall after the study.
* The proportion of patients with preserved renal function (estimated GFR ≥ 60 ml/min) in both treatment arms after the treatment period.
* The proportion of patients with relapse (defines as the reappearance of proteinuria > 3.5 gr/24h and at least 50% increase over the lowest baseline value in at least three consecutive visits in those patients who previously presented a PR or CR) and the time to relapse after the treatment period.
* Serum levels of anti-phospholipase A2 receptor antibodies (anti-PLA2R), before of treatment and at 3, 6, 9, 12, 18 and 24 months of study, in both treatment arms.
* The proportion of patient with drug-related adverse events and serious adverse events.

STUDY POPULATION

Patients with biopsy-proven idiopathic or primary membranous nephropathy with nephrotic proteinuria and normal or slight decrease of renal function will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients are willing and able to read and correctly understand the patient's information sheet and give their consent for participation in the study (by correctly signing and dating the informed consent form document, which has been previously approved by an Ethics Committee/ International Review Board), before initiating any protocol specific selection procedure.
* Patients are able to understand study procedures and to comply with them for the entire length of the study.
* Age older than 18 years.
* Biopsy-proven primary MN. Patients with nephrotic syndrome relapse after remission (either spontaneous or induced by immunosuppression) can be included without a new renal biopsy, provided that they meet all the other inclusion/exclusion criteria.
* Estimated GFR ≥ 45 ml/min/1.73m2 in one measurement performed within the screening period (in the 30 days after informed consent signature).
* Nephrotic-range proteinuria (>4 g/day and not decreasing >50% in the last 6 months) accompanied by hypoalbuminemia ≤ 3, 5 g/dL during the screening period OR patients showing severe or disabling symptoms related to the nephrotic syndrome or severe hypoalbuminemia (<2 g/dL), that can be included before the completion of this 6-month observation period, at the investigator's discretion, independently of proteinuria values.
* Treatment with an ACEI or ARB for at least 2 months before screening (unless intolerance to ACEI/ARB, contraindications to their use or a low blood pressure that could induce side effects at the investigator's discretion) with a controlled blood pressure for at least the last three months (Mean SBP/DBP ≤ 150/90 mmHg in the last three months).
* Negative urine pregnancy test for potentially fertile female.

Exclusion Criteria:

* Diagnosis of secondary causes of membranous nephropathy: malignancy (cancer), systemic infections (which include B and C hepatitis), systemic autoimmune diseases (e.g. Systemic Lupus Erythematosus; SLE) or any other acute or chronic inflammatory disease.
* HIV infection.
* Moderate or severe liver disease (AST and ALT > 2.5x upper range limit and total bilirubin > 1.5 x upper range limit).
* Patients are taking part in any other study with an investigational study and/or are receiving or have received treatment with another investigational drug or intervention (within the first month prior to the signature of the informed consent).
* Suspected or known hypersensitivity, allergy and/or immunogenic reaction history to either rituximab, cyclosporine, tacrolimus, corticosteroids, CYC or any of their ingredients (which include excipients) and of any other drug from the same pharmacotherapeutic group (i.e. calcineurin inhibitors, specific monoclonal antibodies or alkylating agents).
* Previous treatment with corticosteroids in the three months period before screening, or previous treatment with other immunosuppressive agent in the six month period before screening.
* Previous treatment with rituximab or any other biological agent in the two years period before screening.
* Patients who were non-responders to previous immunosuppressants.
* Women with a positive pregnancy test at screening or in lactation period or planning to become pregnant within the next 24 months. Women not willing to use contraceptive methods during the complete study period.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.
* Any other medical unstable, uncontrolled, or severe condition or any other relevant laboratory test finding which, at the investigator's own discretion, could possibly increase the associated risk of the patient's participation in the study.
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete and/or partial remission. | 24 months
  The proportion of patients reaching complete remission, defined as a reduction of proteinuria since baseline level to a value equal or lower than 0.5 g/24 h proteinuria plus stable renal function (eGFR ≥ 45 ml/min/1.73m2) or partial remission, defined as a reduction of proteinuria since baseline level to a value less than 3.5 g/24 h and 50% lower than baseline proteinuria plus stable renal function (eGFR ≥ 45 ml/min/1.73m2) at 24 months of study treatment.

SECONDARY OUTCOMES:
Proportion of patients with limited response | 12, 18, and 24 months
  The proportion of patients with limited response, defined as a reduction of proteinuria since baseline level > 50% but to a value > 3.5g/24 h. at 12, 18 and 24 months of study treatment.
Proportion of patients with increase of baseline serum creatinine ≥ 50% | 12, 18, and 24 months
  The number of patients with an increase ≥ 50% of serum creatinine (SCr) from baseline at 12, 18 and 24 months (end of the follow-up).
Proportions of patients with relapses | 9, 12, 18, and 24 months
  The proportion of patients with relapses (defines as the reappearance of proteinuria > 3.5 gr/24h and at least 50% increase over the lowest baseline value in at least three consecutive visits in those patients who previously presented a PR or CR) and the time to relapse after the treatment period.
Proportion of patients with drug-related adverse events | During all therapy period and until 24 months post-beginning of therapy
  The proportion of patient with drug-related adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: GEMA FERNÁNDEZ-JUÁREZ, MD, Principal Investigator — Hospital Universitario Fundación Alcorcón, Madrid. Spain; JESUS EGIDO, MD, PhD, Principal Investigator — IIS Fundación Jiménez Díaz, Madrid. Spain; MARIAN GOICOCHEA, MD, Principal Investigator — Hospital Universitario Gregorio Marañón, Madrid. Spain; ALFONS SEGARRA, MD, PhD, Principal Investigator — Hospital Universitari Vall d´Hebron, Barcelona. Spain; GUILLERMO MARTÍN, MD, Principal Investigator — Hospital Regional de Málaga, Spain; ILDEFONSO VALERA, MD, Principal Investigator — Hospital Virgen de la Victoria de Málaga. Spain; VIRGINIA CABELLO, MD, Principal Investigator — Hospital Virgen del Rocío, Sevilla. Spain; QUINTANA LUIS, MD, Principal Investigator — Hospital Clinic de Barcelona. Spain; CAO MERCEDES, MD, Principal Investigator — Hospital Universitario de A Coruña. Spain; AVILA ANA, MD, Principal Investigator — Hospital Dr. Peset, Valencia. Spain; ESPINOSA MARIO, MD, Principal Investigator — Hospital Reina Sofía, Córdoba. Spain; MONTSERRAT DIAZ, MD, Principal Investigator — Fundación Puigvert, Barcelona. Spain; BONET JOSÉ, MD, Principal Investigator — Hospital Germans Trias i Pujol, Barcelona. Spain; JUAN RAMÓN GÓMEZ-MARTINO, MD, Principal Investigator — Hospital San Pedro de Alcántara, Cáceres. Spain; RIVAS BEGOÑA, MD, Principal Investigator — Hospital Universitario La Paz; RODRIGUEZ ANTOLINA, MD, Principal Investigator — Hospital Clínico San Carlos, Madrid. Spain; GALEANO CRISTINA, MD, Principal Investigator — Hospital Universitario Ramón y Cajal, Madrid. Spain; RIVERA FRANCISCO, MD, Principal Investigator — Hospital de Ciudad Real. Spain; WETZELS JACK, MD, Principal Investigator — Radboud University Medical Center; JORGE ROJAS, MD, Principal Investigator — IIS Fundación Jiménez Díaz, Madrid. Spain; MARUJA NAVARRO, MD, Principal Investigator — Hospital Germans Trias i Pujol, Barcelona. Spain; ANA ROMERA, MD, Principal Investigator — Hospital de Ciudad Real. Spain; IRENE AGRAZ, MD, Principal Investigator — Hospital Universitari Vall d´Hebron, Barcelona. Spain
Locations (1):
- Hospital 12 de Octubre, Madrid, Spain

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952